CLINICAL TRIAL: NCT00001127
Title: Study of the Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) in a Community-Based, Non-Randomized, Open-Label Trial in Children to Assess Safety and Herd Immunity for the Control of Epidemic Influenza
Brief Title: Study of a Flu Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Aviron LLC (Industry)
Masking: None | Purpose: Prevention
Other Study IDs: DMID 99-021; AV012
Record Dates: First submitted 2000-01-17; First posted 2001-08-31 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2005-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Influenza virus vaccine (CAIV-T)

SUMMARY:
This study tests the safety and effectiveness of a flu vaccine in school children.

School children are usually the first members of a community to come down with the flu, and they often give the flu to their younger siblings, parents, and grandparents. It is hoped that giving school children a flu vaccine can help prevent the spread of the flu to other members of the community.

DETAILED DESCRIPTION:
This is a Phase III trial (an advanced study with a large number of patients). Your child will receive a single dose of flu vaccine, which is given by a nasal spray.

ELIGIBILITY:
Inclusion Criteria:

Your child may be eligible for this study if he/she:

* Is between the ages of 18 months and 18 years, with consent of parent or guardian.
* Is a resident of the Temple-Belton, Texas area.

Exclusion Criteria:

Your child will not be eligible for this study if he/she:

* Has had a fever within 3 days before vaccination.
* Has symptoms of a weakened immune system.
* Has had a wheezing episode within the past 2 weeks.
* Has moderate to severe asthma.
* Is allergic to eggs.
* Needs to take aspirin on a regular basis.
* Has received another vaccine or study drug in the past month.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15000
Dates: Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro A. Piedra, M.D., Houston, Texas, United States